CLINICAL TRIAL: NCT06168760
Title: The Relationship Between Finger-Hand Length And Hand Width With Dexterity In Healthy Individuals
Brief Title: Hand Dexterity and Anthropometric Measurement
Status: Not yet recruiting | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Ömer Faruk ÖZÇELEP, Lecturer, Kirsehir Ahi Evran Universitesi
Other Study IDs: Ahievr
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Anthropometric Measurement; Hand Dexterity
Keywords: anthropometric measurement; hand dexterity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy: Anthropometric measurements of the hand were measured with a digital caliper. Anthropometric measurements were determined as hand length, width and finger lengths, taking into account previous studies. Manual dexterity was evaluated with the 9-Hole Peg Test.
  Interventions: Diagnostic Test: Anthropometric Measurements

INTERVENTIONS:
Diagnostic Test: Anthropometric Measurements — Anthropometric measurements of the hand were measured with a digital caliper. Anthropometric measurements were determined as hand length, width and finger lengths, taking into account previous studies. Manual dexterity was evaluated with the 9-Hole Peg Test.

SUMMARY:
This study aims to investigate the relationship between hand and finger lengths, hand width, and dexterity. The main question it aims to answer is:

1-Is there a relationship between anthropometric measurements of the hand and manual dexterity?

DETAILED DESCRIPTION:
The hand is capable of performing complex specialized tasks that require dexterity, manipulation, and tactile sensitivity.(Polat, 2023) Hand performance on a task is a combination of different skills, including grip muscle strength, movement, tactile feedback, and motor coordination. (Imamura, Rissanen, Kinnunen, & Rintamäki, 1998). To achieve these, the hand is equipped with mechanical and sensory abilities.(Dianat, Haslegrave, & Stedmon, 2012) Dexterity is a motor skill determined by the range of motion of the hands and fingers, as well as the ability to manipulate. It is a combination of reaction time, touch sensation, nerve conduction, grip strength and mobility. While finger dexterity is related to the fine motor skills required to move relatively small objects, manual dexterity includes the gross motor skills required to hold relatively large objects.(Roman et al., 2023) The most common dexterity tests reported in the literature include the Box-Block Test, Purdue Pegboard Test, Jebsen Taylor Test, 9-Hole Peg Test (NHPT), and Roeder Manipulative Ability Test.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers were included if they were 18 years of age or older and did not have any communication disorders

Exclusion Criteria:

* not having undergone any upper extremity surgery and not having a systemic disease

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy Subjects
Sampling Method: Probability Sample
Enrollment: 161 (Estimated)
Dates: Start 2024-03-07 (Estimated); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Hand Dexterity | Baseline and 18 weeks
  Manual dexterity was evaluated with the 9-Hole Peg Test.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided